CLINICAL TRIAL: NCT04042025
Title: A Long-term Follow-up Study of Patients in the Clinical Trials for Spinal Muscular Atrophy Receiving AVXS-101
Brief Title: Long-term Follow-up Study of Patients Receiving Onasemnogene Abeparvovec-xioi
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVXS-101-LT-002; 2019-002611-26 (EudraCT Number); 205305 (Other: JapicCTI); COAV101A12103 (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Spinal Muscular Atrophy Type I; Spinal Muscular Atrophy Type II; Spinal Muscular Atrophy Type III; SMA
Keywords: Gene replacement
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood | interventions — Zolgensma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravenous (IV) & Intrathecal (IT) Onasemnogene Abeparvovec-xioi (Other): Participants received treatment with IV onasemnogene abeparvovec-xioi in an onasemnogene abeparvovec-xioi or received treatment with IT onasemnogene abeparvovec-xioi in an onasemnogene.
  Interventions: Biological: Onasemnogene Abeparvovec-xioi

INTERVENTIONS:
Biological: Onasemnogene Abeparvovec-xioi — Onasemnogene abeparvovec-xioi is a non-replicating recombinant adeno-associated virus serotype 9 containing the human survival motor neuron gene under the control of the cytomegalovirus enhancer/chicken β-actin-hybrid promoter. Onasemnogene abeparvovec-xioi administered as a one-time intravenous (IV) infusion or intrathecal (IT) injection. Dosage determined by participant weight.
  Other Names: Zolgensma

SUMMARY:
This is a long-term follow-up safety and efficacy study of participants in clinical trials for spinal muscular atrophy (SMA) who were treated with onasemnogene abeparvovec-xioi. Participants will roll over from their respective previous (parent) study into this long-term study for continuous monitoring of safety as well as monitoring of continued efficacy and durability of response to onasemnogene abeparvovec-xioi treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any participant with SMA who received onasemnogene abeparvovec-xioi gene replacement therapy in a Novartis Gene Therapies-sponsored clinical study
* Participant/parent/legal guardian willing and able to complete the informed consent process and comply with study procedures and visit schedule

Exclusion Criteria:

* Parent/legal guardian unable or unwilling to participate in the long-term follow-up safety study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Reach Developmental Milestones | Up to 5 years
  Assessed via the developmental milestone checklist, formed of 10 yes/no questions. The developmental milestones are: head control, sitting with support, sitting without support, sitting without support for 30 seconds, hands-and-knees crawling, pulls to stand, standing with assistance, walking with assistance, standing alone and walking alone.
Change From Baseline in Hammersmith Functional Motor Scale - Expanded (HFMSE) Score | Up to 5 years
  The HFMSE was devised for use in children with SMA to give objective information on motor ability and clinical progression. The HFMSE is formed of 33 assessments rated from 0 (unable to perform functional task) to 2 (able to perform functional task unassisted). Higher scores on the total scale of 0-66 indicates higher levels of motor ability.
Number of Participants Who Experience a Clinically Significant Change From Baseline in Pulmonary Assessment Results and Require Ventilatory Support | Up to 15 years
  Participants will receive pulmonary assessments by a pulmonologist or appropriate clinician. Respiratory device data will be reviewed for participants receiving non-invasive ventilatory support.
Number of Participants Who Experience Swallowing Dysfunction and Require Nutritional Support | Up to 5 years
  Assessed via the swallowing function questionnaire, formed of 4 yes/ no questions and 1 body weight question.
Number of Participants Who Experience a Clinically Significant Change from Baseline in Physical Examination Findings | Up to 5 years
  The physical examination includes review of the following systems: head, ears, eyes, nose and throat, lungs/thorax, cardiovascular, abdomen, musculoskeletal, neurologic, dermatologic, lymphatic, and genitourinary. In addition, visual inspection of the spine, back, shoulders, and hips looking for spinal curvature and asymmetry will be carried out. Joints will be assessed for loss of mobility and contractures.
Number of Participants Who Experience a Clinically Significant Change From Baseline in Vital Signs Measurements | Up to 5 years
  Vital sign measurements will include blood pressure, respiratory rate, pulse, axillary temperature, and pulse oximetry.
Change From Baseline in Height Measurements | Up to 5 years
Change From Baseline in Weight Measurements | Up to 5 years
Number of Participants Who Experience a Clinically Significant Change From Baseline in Clinical Laboratory Assessments | Up to 5 years
  Blood samples will be collected for hematology (including complete blood cell count) and chemistry.
Number of Participants Who Experience a Clinically Significant Change From Baseline in Cardiac Assessments | Up to 5 years
  Cardiac assessments will include a 12-lead electrocardiogram, transthoracic echocardiogram and Troponin-I.
Number of Participants Who Experience a Clinically Significant Change From Baseline in Observational Phase Questionnaire Results | Year 6 to Year 15
  The observational phase questionnaire includes 7 yes/no questions. Observation categories include: adverse events, hospitalizations, concomitant medications, ventilatory support and feeding support.
Number of Participants Who Experience at Least One Serious Adverse Event (SAE) | Up to 15 years
  An SAE is defined as any adverse event (appearance of [or worsening of any pre existing]) undesirable sign(s), symptom(s), or medical conditions(s) which meets any one of the following criteria:
  * Fatal
  * Life-threatening
  * Results in persistent or significant disability/incapacity
  * Constitutes a congenital abnormality or birth defect
  * Requires in-patient hospitalization or prolongation of existing hospitalization
  * Is medically significant e.g. defined as an event that jeopardizes the participant or may require medical or surgical intervention to prevent one of the outcomes listed above
Number of Participants Who Experience at Least One Adverse Event of Special Interest (AESI) | Up to 15 years
  An AESI is defined as an AE occurring during any study phase that fulfills one of the following criteria:
  * Hepatotoxicity
  * Thrombotic microangiopathy
  * Cardiac adverse events
  * Dorsal root ganglia toxicity
  * New malignancies
  * New incidence of a neurologic disorder
  * New incidence of an autoimmune disorder
  * New incidence of hematologic disorder
Change From Baseline in Bayley Scales of Infant and Toddler Development | Up to 42 months, 15 days of age
  Third Edition (Bayley-III) to be performed in all patients up to 42 months, 15 days of age.
Change From Baseline in Revised Upper Limb Module (RULM) Score | Up to 5 years
  RULM score is based on a scale from 0 to 37 where lower scores reflect poorer upper limb functional ability.
Change From Baseline in Cogstate Computerized Cognitive Battery Performed in Age 48 Months and Older | Up to 5 years
  The Cogstate Computerized Cognitive Battery consists of the Identification Test (scored 0 (best) to 1.5708 (worst)), the International Shopping List Test (scored 0 (worst) to 999 (best)), the International Shopping List Test-Delayed Recall (scored 0 (worst) to 999 (best)), the One Card Learning Test (scored 0 (worst) to 1.5708 (best)), and the One Back Test (scored 0 (worst) to 1.5708 (best)).
Change From Baseline in Clinical Evaluation of Language Fundamentals Fifth Edition (CELF-5) Performed in All Participants 5 to 21 Years of Age | Up to 5 years
  The CELF-5 Following Directions and Sentence Repetition subtests use scoring that varies based on age, but will be administered to participants 5-21 years of age. The Following Directions subtest will be scored from 0-33 with higher score being more advanced and the Recalling Sentences subtest will be scored from 0-78 with higher score being more advanced.
Change From Baseline in Assessment of Caregiver Experience With Neuromuscular Disease (ACEND) | Up to 5 years
  ACEND score is based on a scale from 1 to 41 where higher scores represent a better caregiver experience
Number of Participants With Concomitant Medications Overall and by Type of Medications | Up to 5 years
Number of Participants With Other SMA Therapies Overall and by Type of Medications | Year 6 to Year 15

CONTACTS AND LOCATIONS:
Overall Officials: Sitra Tauscher-Wisniewski, MD, Study Chair — Novartis Gene Therapies, Inc.
Locations (31):
- United States (18):
  - Stanford University Medical Center, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - John Hopkins Hospital - David M. Rubenstein Child Health Building, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Spectrum Health Hospitals Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Washington Unviersity School of Medicine in Saint Louis, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Clinic for Special Children, Strasburg, Pennsylvania
  - Children's Health Specialty Center Dallas Campus, Dallas, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin, Madison, Madison, Wisconsin
- Sydney Children's Hospital, Randwick, New South Wales, Australia
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - Centre de Référence des Maladies Neuromusculaires, Liège
- Children's Hospital of Eastern Ontario Research Institute, Ottawa, Ontario, Canada
- Hôpital Armand Trousseau, Paris, France
- Italy (4):
  - Instituto Gianninia Gaslini, Genova
  - Universita Degli Studi Di Milano, Milan
  - Istituto Neurologico di Ricerca, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Tokyo Women's Medical University Hospital, Tokyo, Japan
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (2):
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Day JW, Mendell JR, Mercuri E, Finkel RS, Strauss KA, Kleyn A, Tauscher-Wisniewski S, Tukov FF, Reyna SP, Chand DH. Clinical Trial and Postmarketing Safety of Onasemnogene Abeparvovec Therapy. Drug Saf. 2021 Oct;44(10):1109-1119. doi: 10.1007/s40264-021-01107-6. Epub 2021 Aug 12. PMID 34383289